CLINICAL TRIAL: NCT00032487
Title: CSP #465 - Glycemic Control and Complications in Diabetes Mellitus Type 2 (VADT)
Brief Title: Glycemic Control and Complications in Diabetes Mellitus Type 2 (VADT)
Acronym: VADT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Eye Institute (NEI) (NIH); SmithKline Beecham (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 465
Record Dates: First submitted 2002-03-21; First posted 2002-03-22 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: DM; glycemic control; insulin; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin; glimepiride; Rosiglitazone; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard glycemic control (Active Comparator): Standard glycemic control to maintain HbA1c between 8.0-9.0%. Metformin 500 mg Rosiglitazone 4 mg Glimepiride 2 mg Insulin 1 unit 9 lbs
  Interventions: Drug: Insulin; Drug: Glimepiride; Drug: Rosiglitazone; Drug: Metformin
- Intensive glycemic control (Experimental): Intensive glycemic control lower HbA1c below 6.0%. Metformin 500 mg (go up to 2000 mg) Rosiglitazone 4 mg bid Glimepiride 8 mg Insulin 1 unit 9 lbs add one injection to Arm 1
  Interventions: Drug: Insulin; Drug: Glimepiride; Drug: Rosiglitazone; Drug: Metformin

INTERVENTIONS:
Drug: Insulin — Insulin (intermediate or long-lasting) in a.m. 1 unit 9 lbs Arm 1 Insulin (intermediate or long-lasting) in a.m. 1 unit 9 lbs, add one injection of insulin Arm 2
  Other Names: Lente
Drug: Glimepiride — Glimepiride 2 mg Arm 1 Glimepiride 8 mg Arm 2
  Other Names: Amaryl
Drug: Rosiglitazone — Rosiglitazone 4 mg Arm 1 Rosiglitazone 4 mg bid Arm 2
  Other Names: Avandia
Drug: Metformin — Metformin 500 mg (go up to 1000 mg) Arm 1 Metformin 500 mg (go up to 2000 mg) Arm
  Other Names: Glumetza

SUMMARY:
This study is a prospective, 2-arm, randomized controlled trial to determine whether glycemic control, achieved through intensification of treatment, is effective in preventing clinical macrovascular complications in patients with type 2 DM who are no longer responsive to oral agents alone. The study consists of a two-year accrual period and five years of follow-up (7 years total) of 1700 patients across 20 centers. We have powered the study to detect a 21% reduction in the primary event rate. Additional study goals are to determine whether the expenditures, discomfort, and adverse effects associated with intensive intervention are justified in terms of their clinical benefits, considering both macrovascular and microvascular complications.

DETAILED DESCRIPTION:
Primary Hypothesis: Intensive glycemic control reduces major macrovascular morbidity and mortality compared to standard glycemic control in type 2 diabetics who have failed simple therapy.

Secondary Hypotheses: Intensive glycemic control, compared to standard glycemic control, reduces other macrovascular morbidity and total mortality.

Intervention: The intervention is tight glycemic control, aiming at normalization of HbA1c. This will be achieved through stepped care therapy, using all categories of tools available to most diabetologists. These categories include: patient education of diabetes control (e.g. diet, exercise, etc.), oral diabetes medications, and insulin. All drugs to be used are approved. Specific agents will be used within the different classes to promote consistency across sites.

The comparison is standard control, aiming at HbA1c of 8 - 9%. The same agents will be used, but at reduced doses.

The general approach to the stepped care treatment protocol is to treat both groups with the same agents, but at different intensities (doses) (taking into account intolerance/contraindications). The sequence of steps is shown below.

STEP 1: Either Metformin (obese) or Glimepiride (lean)in combination with Rosiglitazone STEP 2: Insulin STEP 3: Increase doses in STEPS 1,2 in the Standard group. Since the Intensive group is already at maximal doses of oral agents, they will intensify insulin and may add Acarbose/Miglitol.

STEP 4: For standard, proceed as in STEP 3 for Intensive; Intensives will use multiple daily injection (MDI) of insulin STEP 5: "Tool Box": Miscellaneous agents, tailored to the individual patient.

Primary Outcomes: Time to one of the following major macrovascular events: myocardial infarction, stroke, new or worsening congestive heart failure, amputation for ischemic gangrene, invasive intervention for coronary artery or peripheral vascular disease, inoperable coronary artery disease, or cardiovascular death.

Secondary Outcomes: Angina, transient ischemic attack, intermittent claudication, critical limb ischemia, and total mortality.

Study Abstract: A quarter of the patients treated by the Department of Veterans Affairs (VA) Health Administration have type 2 diabetes mellitus (DM). The costs of care for the treatment of patients with type 2 DM are extremely high, both in treatment expenditures for the metabolic disorder and for the care of end-organ complications. Although patients initially respond to diet and oral agent treatment, most eventually need insulin to near-normalize their glucose level, as the disease is characterized by progressive loss of insulin secretory capacity.

After several clinical trials in both type 1 and type 2 DM, there is a reasonable certainty that about half of the incidence and rate of progression of indicators of microvascular complications (retinopathy, nephropathy, and neuropathy) can be prevented or delayed by achieving and maintaining near-normalization of glycemic levels. Consequently, there has been a uniform trend in recent guidelines to advise a near-normalization of glycemic levels in both type 1 and type 2 DM. Note, however, that the clinical consequences of microvascular deterioration are dependent not only on glycemic levels but also on the duration of the disease. With the early onset of diabetes typical in type 1 patients, there is sufficient time for development of clinical microvascular complications, and prevention of these complications is a goal of treatment in type 1 diabetics. In contrast, the prevalence of hard clinical endpoints indicative of microangiopathy, such as renal failure or blindness, is very low in patients in whom the disease is diagnosed after the 5th decade, the greatest age of prevalence of patients with type 2 DM in this country. Furthermore, microvascular complications can be minimized by the well-established benefits of blood pressure and lipid control, as well as by therapeutic intervention (photocoagulation, cataract extraction). Since the costs and efforts necessary to reach near-normal levels of glycemia are very high, there is a need to determine the cost/benefit ratios of such expenditures in the population subject to type 2 diabetes, namely patients in their 6th to 8th decades of life.

In contrast with the late and relatively infrequent appearance of clinical endpoints of microangiopathy, macrovascular complications (i.e., coronary heart disease and peripheral vascular disease) are responsible for the overwhelming majority of the mortality, morbidity and treatment costs in the American population of type 2 diabetics, even more so in the older VA diabetic population. In the recently concluded United Kingdom Prospective Diabetes Study (UKPDS) on type 2 DM, macrovascular mortality was 70 times higher than that of microvascular mortality. Intervention studies to determine the effect of rigorous glycemic control on these macrovascular events are inconclusive and contradictory. Intensive treatment in patients who are newly diagnosed has failed to demonstrate a beneficial effect of tight control on cardiovascular complications. The few studies conducted in later stages of the disease (i.e., in patients requiring insulin treatment, alone or in combination with oral agents) have been conflicting and indeterminate.

The decision on intensity of treatment is further compromised by current recommendations to attenuate glycemic control goals, especially when usage of insulin is required, both in patients with the common comorbidities of overweight or preexisting cardiovascular disease, and in those in the later decades of life. These concerns are based on fears that intensive insulin treatment might be associated with weight gain, increased cardiovascular risk factors (hypertriglyceridemia, dyslipidemia, hyperinsulinemia, and insulin resistance), and adverse effects of recurrent hypoglycemic events. The prevalent level of glycemic control in insulin-treated type 2 diabetics is relatively poor, likely due to a combination of practical difficulties and the uncertainties of what are the safe and effective glycemic goals. There is no long-term study currently being done in the high-risk population typical of the patient population in the VA. Before the Department of Veterans Affairs devotes considerable resources to a widespread intervention (a quarter of patients) that may be of little value, and might even be counterproductive, a trial to determine the value of the intervention is mandated. It is expected that CSP #465 will provide the scientific data on which the VA can base clinical treatment of Type II diabetes.

CSP #465 is a prospective, 2-arm, randomized controlled trial to determine whether glycemic control, achieved through intensification of treatment, is effective in preventing clinical macrovascular complications in patients with type 2 DM who are no longer responsive to oral agents alone. The study consists of a two-year accrual period and five years of follow-up (7 years total) of 1700 patients across 20 centers. We have powered the study to detect a 25% reduction in the primary event rate. Additional study goals are to determine whether the expenditures, discomfort, and adverse effects associated with intensive intervention are justified in terms of their clinical benefits, considering both macrovascular and microvascular complications.

Main Manuscript:Duckworth W, Abraira C, Moritz T, Reda D, Emanuele N et al., VADT investigators: Glucose Control and Complications in the VA Diabetes Trial (VADT). N Eng J of Med 360:129-139, 2009.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 DM who are no longer responsive to maximum dose of one or more oral agents.

Exclusion Criteria:

* Angina pectoris, Canadian Class I-II,
* congestive heart failure, Class III-IV,
* stroke, incapacitating or in last 6 months,
* Myocardial infarction (MI) or invasive cardiovascular procedure within the past six months,
* ongoing diabetic gangrene,
* BMI > 40,
* hemoglobinopathy that interferes with A1c monitoring,
* serum creatinine > 1.6 mg/dL,
* fasting C-peptide < 0.21 pmol/ml,
* Alanine Amino Transaminase (ALT) > 3 times normal or serum bilirubin > 1.9 mg/dL,
* malignancy or noncardiac life-threatening diseases making life expectancy < 5 years,
* autonomic neuropathy,
* symptomatic pancreatic insufficiency (endocrine or exocrine),
* recurrent seizures within the past year,
* hypopituitarism,
* pregnancy, lactation, or planning a pregnancy,
* active psychosis or substance abuse,
* lack of access to a person who can assist or be called in an emergency,
* underlying conditions that in the site PI's judgment may prevent adherence to protocol,
* current participation in another clinical trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1791 (Actual)
Dates: Start 2000-12-01 (Actual); Primary Completion 2008-05-30 (Actual); Study Completion 2008-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Abraira, MD, Study Chair — Miami VA Healthcare System, Miami, FL; William Duckworth, MD, Study Chair — Phoenix VA Health Care System, Phoenix, AZ
Locations (21):
- United States (20):
  - Carl T. Hayden VA Medical Center, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Tucson, Arizona
  - VA Central California Health Care System, Fresno, Fresno, California
  - VA Medical Center, Long Beach, Long Beach, California
  - VA San Diego Healthcare System, San Diego, San Diego, California
  - Miami VA Healthcare System, Miami, FL, Miami, Florida
  - Edward Hines, Jr. VA Hospital, Hines, Illinois
  - Richard Roudebush VA Medical Center, Indianapolis, Indianapolis, Indiana
  - VA Medical Center, Lexington, Lexington, Kentucky
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - VA Medical Center, Omaha, Omaha, Nebraska
  - VA New Jersey Health Care System, East Orange, East Orange, New Jersey
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - Ralph H Johnson VA Medical Center, Charleston, Charleston, South Carolina
  - VA Medical Center, Nashville, Tennessee
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA South Texas Health Care System, San Antonio, San Antonio, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - VA Medical Center, Salem VA, Salem, Virginia
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington
- VA Medical Center, San Juan, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duckworth W, Abraira C, Moritz T, Reda D, Emanuele N, Reaven PD, Zieve FJ, Marks J, Davis SN, Hayward R, Warren SR, Goldman S, McCarren M, Vitek ME, Henderson WG, Huang GD; VADT Investigators. Glucose control and vascular complications in veterans with type 2 diabetes. N Engl J Med. 2009 Jan 8;360(2):129-39. doi: 10.1056/NEJMoa0808431. Epub 2008 Dec 17. PMID 19092145
- [Result] Moritz T, Duckworth W, Abraira C. Veterans Affairs diabetes trial--corrections. N Engl J Med. 2009 Sep 3;361(10):1024-5. doi: 10.1056/NEJMc096250. No abstract available. PMID 19726779
- [Result] Emanuele N, Moritz T, Klein R, Davis MD, Glander K, Khanna A, Thottapurathu L, Bahn G, Duckworth W, Abraira C; Veterans Affairs Diabetes Trial Study Group. Ethnicity, race, and clinically significant macular edema in the Veterans Affairs Diabetes Trial (VADT). Diabetes Res Clin Pract. 2009 Nov;86(2):104-10. doi: 10.1016/j.diabres.2009.08.001. Epub 2009 Aug 31. PMID 19720420
- [Result] Control Group; Turnbull FM, Abraira C, Anderson RJ, Byington RP, Chalmers JP, Duckworth WC, Evans GW, Gerstein HC, Holman RR, Moritz TE, Neal BC, Ninomiya T, Patel AA, Paul SK, Travert F, Woodward M. Intensive glucose control and macrovascular outcomes in type 2 diabetes. Diabetologia. 2009 Nov;52(11):2288-98. doi: 10.1007/s00125-009-1470-0. Epub 2009 Aug 5. PMID 19655124
- [Result] Abraira C, Duckworth WC, Moritz T; VADT Group. Glycaemic separation and risk factor control in the Veterans Affairs Diabetes Trial: an interim report. Diabetes Obes Metab. 2009 Feb;11(2):150-6. doi: 10.1111/j.1463-1326.2008.00933.x. Epub 2008 Jul 29. PMID 18671796
- [Result] Emanuele N, Klein R, Moritz T, Davis MD, Glander K, Anderson R, Reda D, Duckworth W, Abraira C; VADT Study Group. Comparison of dilated fundus examinations with seven-field stereo fundus photographs in the Veterans Affairs Diabetes Trial. J Diabetes Complications. 2009 Sep-Oct;23(5):323-9. doi: 10.1016/j.jdiacomp.2008.02.010. Epub 2008 Apr 11. PMID 18406632
- [Result] Meyers CD, McCarren M, Wong ND, Abraira C, Duckworth WC, Kashyap ML; VADT Investigators. Baseline achievement of lipid goals and usage of lipid medications in patients with diabetes mellitus (from the Veterans Affairs Diabetes Trial). Am J Cardiol. 2006 Jul 1;98(1):63-5. doi: 10.1016/j.amjcard.2006.01.061. Epub 2006 May 4. PMID 16784922
- [Result] Duckworth WC, McCarren M, Abraira C; VADT Investigators. Control of cardiovascular risk factors in the Veterans Affairs Diabetes Trial in advanced type 2 diabetes. Endocr Pract. 2006 Jan-Feb;12 Suppl 1:85-8. doi: 10.4158/EP.12.S1.85. PMID 16627388
- [Result] Kirkman MS, McCarren M, Shah J, Duckworth W, Abraira C; VADT Study Group. The association between metabolic control and prevalent macrovascular disease in Type 2 diabetes: the VA Cooperative Study in diabetes. J Diabetes Complications. 2006 Mar-Apr;20(2):75-80. doi: 10.1016/j.jdiacomp.2005.06.013. PMID 16504835
- [Result] Emanuele N, Sacks J, Klein R, Reda D, Anderson R, Duckworth W, Abraira C; Veterans Affairs Diabetes Trial Group. Ethnicity, race, and baseline retinopathy correlates in the veterans affairs diabetes trial. Diabetes Care. 2005 Aug;28(8):1954-8. doi: 10.2337/diacare.28.8.1954. PMID 16043738
- [Result] Abraira C, Duckworth W, McCarren M, Emanuele N, Arca D, Reda D, Henderson W; VA Cooperative Study of Glycemic Control and Complications in Diabetes Mellitus Type 2. Design of the cooperative study on glycemic control and complications in diabetes mellitus type 2: Veterans Affairs Diabetes Trial. J Diabetes Complications. 2003 Nov-Dec;17(6):314-22. doi: 10.1016/s1056-8727(02)00277-5. PMID 14583175
- [Result] Duckworth WC, McCarren M, Abraira C; VA Diabetes Trial. Glucose control and cardiovascular complications: the VA Diabetes Trial. Diabetes Care. 2001 May;24(5):942-5. doi: 10.2337/diacare.24.5.942. No abstract available. PMID 11347758
- [Result] Anderson RJ, Bahn GD, Moritz TE, Kaufman D, Abraira C, Duckworth W; VADT Study Group. Blood pressure and cardiovascular disease risk in the Veterans Affairs Diabetes Trial. Diabetes Care. 2011 Jan;34(1):34-8. doi: 10.2337/dc10-1420. Epub 2010 Nov 8. PMID 21059830
- [Result] Agrawal L, Azad N, Emanuele NV, Bahn GD, Kaufman DG, Moritz TE, Duckworth WC, Abraira C; Veterans Affairs Diabetes Trial (VADT) Study Group. Observation on renal outcomes in the Veterans Affairs Diabetes Trial. Diabetes Care. 2011 Sep;34(9):2090-4. doi: 10.2337/dc11-0175. Epub 2011 Jul 20. PMID 21775749
- [Derived] Zhou JJ, Koska J, Bahn G, Reaven P. Fasting Glucose Variation Predicts Microvascular Risk in ACCORD and VADT. J Clin Endocrinol Metab. 2021 Mar 25;106(4):1150-1162. doi: 10.1210/clinem/dgaa941. PMID 33367811
- [Derived] Reaven PD, Emanuele NV, Wiitala WL, Bahn GD, Reda DJ, McCarren M, Duckworth WC, Hayward RA; VADT Investigators. Intensive Glucose Control in Patients with Type 2 Diabetes - 15-Year Follow-up. N Engl J Med. 2019 Jun 6;380(23):2215-2224. doi: 10.1056/NEJMoa1806802. PMID 31167051
- [Derived] Davis SN, Duckworth W, Emanuele N, Hayward RA, Wiitala WL, Thottapurathu L, Reda DJ, Reaven PD; Investigators of the Veterans Affairs Diabetes Trial. Effects of Severe Hypoglycemia on Cardiovascular Outcomes and Death in the Veterans Affairs Diabetes Trial. Diabetes Care. 2019 Jan;42(1):157-163. doi: 10.2337/dc18-1144. Epub 2018 Nov 19. PMID 30455335
- [Derived] Azad N, Bahn GD, Emanuele NV, Agrawal L, Ge L, Reda D, Klein R, Reaven PD, Hayward R; VADT Study Group. Association of Blood Glucose Control and Lipids With Diabetic Retinopathy in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2016 May;39(5):816-22. doi: 10.2337/dc15-1897. Epub 2016 Mar 22. PMID 27006510
- [Derived] Saremi A, Bahn GD, Reaven PD; Veterans Affairs Diabetes Trial (VADT). A Link Between Hypoglycemia and Progression of Atherosclerosis in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2016 Mar;39(3):448-54. doi: 10.2337/dc15-2107. Epub 2016 Jan 19. PMID 26786575
- [Derived] Hayward RA, Reaven PD, Wiitala WL, Bahn GD, Reda DJ, Ge L, McCarren M, Duckworth WC, Emanuele NV; VADT Investigators. Follow-up of glycemic control and cardiovascular outcomes in type 2 diabetes. N Engl J Med. 2015 Jun 4;372(23):2197-206. doi: 10.1056/NEJMoa1414266. PMID 26039600
- [Derived] Saremi A, Schwenke DC, Bahn G, Ge L, Emanuele N, Reaven PD; VADT Investigators. The effect of intensive glucose lowering therapy among major racial/ethnic groups in the Veterans Affairs Diabetes Trial. Metabolism. 2015 Feb;64(2):218-25. doi: 10.1016/j.metabol.2014.10.010. Epub 2014 Oct 17. PMID 25456099
- [Derived] Anderson RJ, Bahn GD, Emanuele NV, Marks JB, Duckworth WC; VADT Study Group. Blood pressure and pulse pressure effects on renal outcomes in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2014 Oct;37(10):2782-8. doi: 10.2337/dc14-0284. Epub 2014 Jul 21. PMID 25048382
- [Derived] Koska J, Saremi A, Bahn G, Yamashita S, Reaven PD; Veterans Affairs Diabetes Trial Investigators. The effect of intensive glucose lowering on lipoprotein particle profiles and inflammatory markers in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2013 Aug;36(8):2408-14. doi: 10.2337/dc12-2082. Epub 2013 Mar 27. PMID 23536583
- [Derived] Saremi A, Moritz TE, Anderson RJ, Abraira C, Duckworth WC, Reaven PD; Veterans Affairs Diabetes Trial (VADT). Rates and determinants of coronary and abdominal aortic artery calcium progression in the Veterans Affairs Diabetes Trial (VADT). Diabetes Care. 2010 Dec;33(12):2642-7. doi: 10.2337/dc10-1388. Epub 2010 Aug 31. PMID 20807873
- [Derived] Meier M, Hummel M. Cardiovascular disease and intensive glucose control in type 2 diabetes mellitus: moving practice toward evidence-based strategies. Vasc Health Risk Manag. 2009;5:859-71. doi: 10.2147/vhrm.s4808. Epub 2009 Nov 2. PMID 19898642

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty Veterans Affairs Medical Centers (VAMCs) were selected to participate in this cooperative study. The recruitment period was from 12/01/00 to 05/31/03.
Pre-assignment Details: A patient had to meet all the screening criteria for eligibility and had to sign a consent form with blood samples and meet all entry criteria for pre-randomization testing. Once the patient was deemed appropriate for the study, Hines completed the randomization assignment.
Period: Overall Study
Arm/Group | Standard Glycemic Control | Intensive Glycemic Control
Started | 899 | 892
Completed | 760 | 772
Not Completed | 139 | 120
Not completed — Withdrawal by Subject | 67 | 43
Not completed — Adverse Event | 3 | 7
Not completed — Lost to Follow-up | 57 | 58
Not completed — Had other reason | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Arm 1/Standard Glycemic Control: Standard glycemic control to maintain HbA1c between 8.0-9.0%. Metformin 500 mg Rosiglitazone 4 mg Glimepiride 2 mg Insulin 1 unit 9 lbs
- Arm 2/Intensive Glycemic Control: Intensive glycemic control lower HbA1c below 6.0%. Metformin 500 mg (go up to 2000 mg) Rosiglitazone 4 mg bid Glimepiride 8 mg Insulin 1 unit 9 lbs add one injection to Standard glycemic control
- Total: Total of all reporting groups
Arm/Group | Arm 1/Standard Glycemic Control | Arm 2/Intensive Glycemic Control | Total
Number analyzed (Participants) | 899 | 892 | 1791
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 606 | 612 | 1218
  >=65 years | 293 | 280 | 573
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (9.0) | 60.5 (9.0) | 60.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 873 | 866 | 1739
Region of Enrollment [Number; unit: participants]
  United States | 899 | 892 | 1791

OUTCOME MEASURES:

1. Primary Outcome: Primary Major Macrovascular Events
Description: Myocardial infarction (MI), intervention for coronary artery or Peripheral Vascular Disease (PVD), severe inoperable Coronary Artery Disease (CAD), new or worsening Congestive Heart Failure (CHF), stroke, Cardiovascular (CV) death, or amputation for ischemic gangrene.
Time Frame: Post baseline time to the first major macrovascular event up to 82 months
Measure: Number; unit: participants
Groups:
- Arm 1: Standard glycemic control to maintain HbA1c between 8.0-9.0%. Metformin 500 mg Rosiglitazone 4 mg Glimepiride 2 mg Insulin 1 unit 9 lbs
- Arm 2: Intensive glycemic control lower HbA1c below 6.0%. Metformin 500 mg (go up to 2000 mg) Rosiglitazone 4 mg bid Glimepiride 8 mg Insulin 1 unit 9 lbs add one injection to Arm 1
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 899 | 892
participants | 264 | 235
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2; It was hypothesized 21% reduction in intensive glycemic control group compared to standard control group on primary cardiovascular composite outcomes; Test type: Non-Inferiority or Equivalence — The statistical analysis tested was for equivalence. We assumed 86% power with 21% of effect size and the sample size 1700 with 5% drop out rate; p < 0.05, Log Rank; Cox Proportional Hazard = 0.79, 95% CI 2-sided [.79 to .99]

2. Secondary Outcome: Secondary Endpoint
Description: New or worsening angina, new transient ischemic attack (TIA), new intermittent claudication or critical limb ischemia with Doppler evidence or total mortality.
Time Frame: Post baseline time to first event up to 82 months
Measure: Number; unit: participants
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 899 | 892
participants | 283 | 312

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a 82-month period.
Description: Adverse events were reported by staff at visits or the patient between visits. Staff submitted an Adverse event report, using the FDA Form 3500, for each patient with a severe or unexpected reaction that may reasonably be treatment-related. Reports were screened by the research pharmacist and Study Co-Chairs.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 144/899 | 197/892
Other Adverse Events (participants affected / at risk) | 730/899 | 675/892
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=899) | Arm 2 (N=892)
Infections and infestations (Infections and infestations) | 81 (81) | 71 (71)
Cardiac disorders (Cardiac disorders) | 36 (36) | 40 (40)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 20 (20) | 38 (38)
Gastrointestinal disorders (Gastrointestinal disorders) | 40 (40) | 37 (37)
General Disorders (General disorders) | 32 (32) | 36 (36)
Nervous System Disorders (Nervous system disorders) | 29 (29) | 36 (36)
Respiratory, thoracic and mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 25 (25) | 36 (36)
Surgical and Medical Procedures (Surgical and medical procedures) | 37 (37) | 33 (33)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 25 (25) | 27 (27)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 31 (31) | 26 (26)
Renal and Urinary Disorders (Renal and urinary disorders) | 25 (25) | 26 (26)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 (25) | 23 (23)
Investigations (Investigations) | 22 (22) | 22 (22)
Vascular Disorders (Vascular disorders) | 22 (22) | 20 (20)
Blood and lymphatic Disorders (Blood and lymphatic system disorders) | 12 (12) | 15 (15)
Skin and subcutaneous tissue Disorders (Skin and subcutaneous tissue disorders) | 4 (4) | 12 (12)
Hepatobiliary Disorders (Hepatobiliary disorders) | 6 (6) | 9 (9)
Psychiatric Disorders (Psychiatric disorders) | 14 (14) | 7 (7)
Reproductive system and brest Disorders (Reproductive system and breast disorders) | 2 (2) | 6 (6)
Congenital, familial and genetic Disorders (Congenital, familial and genetic disorders) | 2 (2) | 4 (4)
Eye Disorders (Eye disorders) | 6 (6) | 2 (2)
Endocrine Disorders (Endocrine disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=899) | Arm 2 (N=892)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 493 (493) | 480 (480)
Infections (Infections and infestations) | 385 (385) | 354 (354)
General Disorders (General disorders) | 315 (315) | 290 (290)
Nervous system (Nervous system disorders) | 318 (318) | 283 (283)
Gastrointestinal Disorders (Gastrointestinal disorders) | 288 (288) | 289 (289)
Injury (Injury, poisoning and procedural complications) | 235 (235) | 227 (227)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 227 (227) | 218 (218)
Skin (Skin and subcutaneous tissue disorders) | 214 (214) | 206 (206)
Investigations (Investigations) | 167 (167) | 174 (174)
Eye Disorders (Eye disorders) | 185 (185) | 183 (183)
Psychiatric (Psychiatric disorders) | 175 (175) | 166 (166)
Renal (Renal and urinary disorders) | 138 (138) | 158 (158)
Metabolism (Metabolism and nutrition disorders) | 115 (115) | 132 (132)
Vascular (Vascular disorders) | 115 (115) | 90 (90)
Surgical (Surgical and medical procedures) | 77 (77) | 89 (89)
Cardiac Disorders (Cardiac disorders) | 69 (69) | 62 (62)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 78 (78) | 64 (64)
Blood (Blood and lymphatic system disorders) | 67 (67) | 87 (87)
Reproductive (Reproductive system and breast disorders) | 82 (82) | 62 (62)
Immune (Immune system disorders) | 67 (67) | 58 (58)
Ear (Ear and labyrinth disorders) | 61 (61) | 52 (52)

LIMITATIONS AND CAVEATS:
Our study had several limitations. Since we were studying veterans, the patients were predominantly men, and extrapolation of our findings to women must be done with caution.Changes in therapeutic agents have occurred since the design of our protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes